CLINICAL TRIAL: NCT02184364
Title: Double-blind Dose/Response Study Comparing Klimadynon® With Conjugated Oestrogens in Women Suffering From Menopausal Complaints
Brief Title: Klimadynon® in Comparison to Conjugated Oestrogens in Women Suffering From Menopausal Complaints
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 563.1
Record Dates: First submitted 2014-07-08; First posted 2014-07-09 (Estimated); Last update posted 2014-07-14 (Estimated); Status verified 2014-07

CONDITIONS: Menopause
MeSH Terms: interventions — Klimadynon; Estrogens, Conjugated (USP)

ARMS (5):
- Low dose of Klimadynon® (Experimental)
  Interventions: Drug: Low dose of Klimadynon®
- Medium dose of Klimadynon® (Experimental)
  Interventions: Drug: Medium dose of Klimadynon®
- High dose of Klimadynon® (Experimental)
  Interventions: Drug: High dose of Klimadynon®
- Oestrofeminal® (Active Comparator)
  Interventions: Drug: Oestrofeminal®
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Low dose of Klimadynon®
  Arms: Low dose of Klimadynon®
Drug: Medium dose of Klimadynon®
  Arms: Medium dose of Klimadynon®
Drug: High dose of Klimadynon®
  Arms: High dose of Klimadynon®
Drug: Oestrofeminal®
  Arms: Oestrofeminal®
Drug: Placebo
  Arms: Placebo

SUMMARY:
To investigate, relative to placebo and conjugated oestrogens, the efficacy, safety and tolerability of a 12 weeks peroral treatment twice daily with a cimicifuga racemosa extract corresponding to 20 mg, 75 mg or 150 mg plant material on menopause-related neurovegetative and mental complaints

ELIGIBILITY:
Inclusion Criteria:

* Only postmenopausal (amenorrhea for 6 months at least) women may be enrolled in the study
* Women after ovariectomy may also be enrolled if surgery was carried out at least 6 months prior to the enrollment. Only women between the age of 40 and 60 may be included
* 2 weeks (control -1, week -2, day -14) before the beginning of the treatment the following hormone values must have been analyzed:

  * estradiol-17ß ≤ 0.15 nmol/l corresponding to ≤ 40 pg/ml and follicle stimulating hormone (FSH) ≥ 25 milliunits per milliliter (mU/ml)
  * These hormone analyses must be carried out at the competent local laboratory
* In addition to other menopausal complaints the women must have hot flushes / outbreaks of sweating:

  * Diary: During the "run-in period" daily ≥ 3 hot flushes / outbreaks of sweating
  * Modified Menopause Rating Scale, 1st item twofold (week -2 and 0) ≥ 0.3
* A sum score taken twice from the modified (only items 1 - 6) Menopause Rating Scale within 2 weeks (week - 1 and 0) before the beginning of treatment must be ≥ 1.7
* In case of a pretreatment with estrogen a wash-out phase of 6 weeks is necessary in case of oral or transdermal administration. After the 4th week of wash-out the patient may be included in the "run-in period"

Exclusion Criteria:

* General criteria for exclusion:

  * Non-responder (= no therapeutic success) under a pretreatment with estrogen
  * Amenorrhea for < 6 months
  * In case of an estrogen pretreatment last menstruation (menopause) > 3 years earlier
  * Sum score of the modified Menopause Rating Scale (items 1 - 6) during the "run-in period" twice (week -2 and 0) < 1.7
  * No hot flushes / outbreaks of sweating (see Inclusion criteria)
  * At one of the appointments of the "run-in period" (week -2 and 0) more than one question of items 1 - 6 of the modified Menopause Rating Scale (MMRS) not answered
  * During the "run-in period" at the appointment week -2: estradiol-17ß > 40 pg/ml corresponding to > 0.15 nmol/l and FSH < 25 mU/ml
  * Condition after hysterectomy
  * Simultaneous ingestion of estrogen-containing products in addition to the test products
  * Any addition ingestion of psychotropic drugs, antidepressants and sleeping aids (hypnotics / sedatives)
  * Treatment with another study drug in the 2 months preceding the beginning of the study
  * Considerable overweight (exceeding the target body weight [height in cm minus 100] by more than 30%)
  * Poor general condition
  * Alcohol or drug abuse
  * Poor compliance
* Exclusion criteria based on conjugated estrogens or medroxyprogesterone:

  * Any contraindication for estrogen
  * Unresolved genital bleeding
  * Suspicion / existence of estrogen-dependent mammary carcinoma (mammography and/or endometrial carcinoma)
  * Endometriosis
  * Endometrial hyperplasia (including hyperplastic polypoid endometrium, which has not yet reached the stage of a glandular cystic hyperplasia)
  * Thickness of endometrium > 5 mm
  * Existing thromboembolism or thromboembolism in the past
  * Phlebitis in the past 2 years or actually existing
  * Acute or chronic hepatic lesion (aspartate transaminase and/or alanine transaminase and/or gamma glutamyl transferase twice the normal range)
  * Metabolic disorders of bile pigments (Dubin-Johnson's syndrome, Rotor syndrome, pregnancy icterus with/without pruritus in previous pregnancy)
  * Sickle cell anemia
  * Clinically relevant hypertriglyceridemia or hypercholesterolemia
  * Heart attack in the past
  * Severe varicosis
  * Known sensitivity to medroxyprogesterone
  * Case history of anaphylactic reaction
  * Any neoplasm at the genitals
  * Case history of antidepressant treatment
  * Diabetes mellitus with or without treatment

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 161 (Actual)
Dates: Start 1998-11; Primary Completion 2000-09 (Actual)

PRIMARY OUTCOMES:
Change of score in menopause-related symptom categories of the modified menopausal rating scale (MRS) | baseline, week 12

SECONDARY OUTCOMES:
Change of score of MRS items 7-10 and items 1-10 | baseline, week 12
Change of menopause index according to Kupperman | Baseline up to day 98
  a 4 point numerical scale rating of 11 weighted menopause-related symptom complexes
Changes in daily frequency of menopausal lead symptoms | Up to day 105
  diary information
Changes from baseline in serum concentration of oestradiol-17ß | Up to day 98
Changes from baseline in serum concentration of FSH | Up to day 98
Changes from baseline in serum concentration of luteinising hormone | Up to day 98
Changes from baseline in serum concentration of osteocalcin | Up to day 98
Changes from baseline in serum concentration of ß-CrossLaps | Up to day 98
Changes from baseline in serum concentration of bone specific alkaline phosphatase | Up to day 98
Changes from baseline in serum concentration of cholesterol | Up to day 98
Changes from baseline in serum concentration of high density lipoproteins | Up to day 98
Changes from baseline in serum concentration of low density lipoproteins | Up to day 98
Changes from baseline in serum concentration of triglycerides | Up to day 98
Changes from baseline in serum concentration of glucose | Up to day 98
Changes from baseline in maturity index of the vaginal epithelium | Baseline, day 84
Assessment of global efficacy evaluated by patient and investigator on a 4-point rating scale | At day 98
Changes from baseline in thickness of endometrium | Baseline, day 84
  measured in millimeters, assessed by transvaginal ultrasonography
Diary information regarding frequency, duration and intensity of vaginal bleeding on treatment | Up to day 105
Changes from baseline for mammography/ ultrasonography assessment of the breasts | Baseline, day 98
Changes from baseline in vital signs (blood pressure, heart rate) | Baseline up to day 98
Number of patients with adverse events | Up to day 105
Changes from baseline in clinical laboratory including coagulation parameters | Baseline, day 56, day 98
Assessment for incidence of withdrawal bleeding upon peroral gestagen administration | At day 105
Assessment of global tolerability evaluated by patient and investigator (4-point rating scale) | At day 98
Change in scores of major climacteric complaints (MRS items 1, 4, 9, 10) | baseline, week 12
Change in scores of somatic complaints (MRS items 1, 2, 8, 9, 10) | baseline, week 12
Changes from baseline in body weight | Baseline up to day 98